CLINICAL TRIAL: NCT02246543
Title: Whey Protein Study - Identification of Sustainable Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2/033/13; 132033 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2014-09-15; First posted 2014-09-22 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Satiety
Keywords: Appetite; Gut Hormones; Protein; Energy Density; Gastric Emptying

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment 1 - Control (Placebo Comparator): Water, Toast & Egg (Yolk only) + 0.1g 13C Octanoic Acid
  Interventions: Dietary Supplement: Control
- Treatment 2 - HPL (Active Comparator): High Protein Smoothie (Liquid): 30% protein; 30% fat and 40% CHO + 0.1g 13C Octanoic Acid
  Interventions: Dietary Supplement: HPL
- Treatment 3 - LPL (Active Comparator): Low Protein Smoothie (Liquid): 15% protein; 30% fat and 55% CHO + 0.1g 13C Octanoic Acid
  Interventions: Dietary Supplement: LPL
- Treatment 4 - HPS (Active Comparator): High Protein Milk Jelly (Solid): 30% protein; 30% fat and 40% CHO + 0.1g 13C Octanoic Acid
  Interventions: Dietary Supplement: HPS
- Treatment 5 - LPS (Active Comparator): Low Protein Milk Jelly (Solid): 15% protein; 30% fat and 55% CHO + 0.1g 13C Octanoic Acid
  Interventions: Dietary Supplement: LPS

INTERVENTIONS:
Dietary Supplement: Control — Water, Toast & Egg (Yolk only) + 0.1g 13C Octanoic Acid
  Arms: Treatment 1 - Control
Dietary Supplement: HPL — High Protein Smoothie (Liquid): 30% protein; 30% fat and 40% CHO + 0.1g 13C Octanoic Acid
  Arms: Treatment 2 - HPL
Dietary Supplement: LPL — Low Protein Smoothie (Liquid): 15% protein; 30% fat and 55% CHO + 0.1g 13C Octanoic Acid
  Arms: Treatment 3 - LPL
Dietary Supplement: HPS — High Protein Milk Jelly (Solid): 30% protein; 30% fat and 40% CHO + 0.1g 13C Octanoic Acid
  Arms: Treatment 4 - HPS
Dietary Supplement: LPS — Low Protein Milk Jelly (Solid): 15% protein; 30% fat and 55% CHO + 0.1g 13C Octanoic Acid
  Arms: Treatment 5 - LPS

SUMMARY:
This study will have the primary aim to investigate within-day changes in appetite after consumption of high-protein (HP, 30% of calories) and normal, or low, protein (LP, 15% of calories) whey protein meal, in solid and liquid form, on appetite and ad libitum food intake. Secondary objective will be to assess the statistical relationship between plasma concentrations of gut hormones and visual analogue scales (subjective hunger and fullness) and transit time.

In order to investigate the interaction of food structure and protein content on appetite, this requires, in practice, either a differing amount (g) or calorie (kJ) load as a function of energy density (defined as kJ/100g). Delivering the test meal as a solid and liquid form gives an easy solution to achieve this manipulation without compromising the nutritional profile. Following on from this decision, it is easier to produce different preloads using whey protein (rather than meat protein), since it is easily incorporated into test meals.

DETAILED DESCRIPTION:
A randomized crossover design in 10 overweight/obese (BMI 26-40) men and 10 lean men (BMI 18.5-25). The control will be water. Each subject will attend the HNU on six separate occasions. The five test meal challenges will involve subjects attending the Human Nutrition Unit (HNU) in the morning, after an overnight fast. The total time of test meal visits will be approximately 4½hours. They will be provided with a standardised meal, after which blood samples will be collected for the first 2hrs. The following five treatments will be tested:

Treatment 1 Control - Water + Egg Yolk Mixture + 13C Octanoic Acid Treatment 2 HPL (High Protein Liquid): 30% protein; 30% fat and 40% carbohydrate (CHO) Treatment 3 LPL (Low Protein Liquid): 15% protein; 30% fat and 55% CHO Treatment 4 HPS (High Protein Solid): 30% protein; 30% fat and 40% CHO Treatment 5 LPS (Low Protein Solid): 15% protein; 30% fat and 55% CHO Test meals will be of fixed nutritional composition for all participants. The liquid meal will be a milk/fruit smoothie mixture and the 'solid' will be in a milk jelly (set) form.

Ad libitum pasta meal: 15% protein; 30% fat and 55% CHO as a homogenous mix and energy density of around 400kJ/100g - served in excess as a individual 600g portion to 'help-yourself'.

Subjective average appetite will be measured (every 30 min by visual analogue scales) over 4hr and ad libitum food intake will measured 4hr after treatment consumption. Ad libitum lunch will be a homogenous pasta meal with tomato sauce and a bottle of water. Blood samples will be collected every 10 min for the first half hour, every 15 min for the second half hour and every 30mins subsequently. The breath gastric emptying measurement will be assessed using the 13Carbon (13C) Octanoic Acid stable isotopic technique19. This involves mixing the tracer into food and taking breath samples and measured by isotope ratio mass spectrometry. 13C Octanoic acid is a medium chain fatty acid which is rapidly absorbed in the duodenum and metabolised in the liver. Following oxidation, the resulting Carbon Dioxide (CO2) is excreted into breath (12 samples will be collected during the 4hr test day).

ELIGIBILITY:
Inclusion Criteria:

* BMI = 18.5-40kg/m2

Exclusion Criteria:

* Diabetes
* Severe gastrointestinal disorders
* Kidney disease
* Thromboembolic or coagulation disease
* Hepatic disease
* Alcohol or any other substance abuse
* Gout
* Eating disorders
* Food allergy
* Unregulated thyroid disease
* Psychiatric disorders (including severe depression, lithium treatment, schizophrenia, severe behavioural disorders)
* Vegetarians & Vegans

Medication Exclusion Criteria:

* Orlistat (Xenical)
* Oral antidiabetics, insulin
* Rimonabant (Acomplia)
* Digoxin, anti-arrhythmics
* Sibutramine (Reductil)
* Tricyclic antidepressants, neuroleptics

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Changes in postprandial biomarkers of satiety as measured by gut-related hormones | On each test day blood samples are collected every 10 min for the first half hour, every 15 min for the second half hour and every 30mins subsequently. (Eight samples are therefore collected for 2hours at T0, T10, T20, T30, T45, T60, T90 and T120mins)
  The biomarkers to be measured on the Luminex system are Ghrelin (active), Glucagon-like peptide (GLP1), Peptide YY (PYY), Amylin, Leptin & Insulin
  Biomarkers of Cardiovascular Disease (CVD) risk including total cholesterol, Low Density Lipoprotein Cholesterol (LDL), High Density Lipoprotein (HDL), triglycerides, nonesterified fatty acids (NEFA) will also be measured along with assessment of peripheral glycaemic control, fasting glucose, area under the curve combined with insulin data.

SECONDARY OUTCOMES:
Changes in postprandial gastric emptying, measured using breath samples | On each test day samples are collected every 15mins for the first 2½hrs then every 30mins for the last ½hr. Therefore samples are collected for a total of 3hours at T0, T15, T30, T45, T60, T75, T90, T105, T120, T135, T150 and T180mins.
  This is assessed using the 13C Octanoic Acid stable isotopic technique. A tracer is mixed into food and breath samples are collected which are analysed by isotope ratio mass spectrometry. 13C Octanoic acid is a medium chain fatty acid which is rapidly absorbed in the duodenum and metabolised in the liver. Following oxidation, the resulting CO2 is excreted into breath (12 samples will be collected during the 4hr test day).

OTHER OUTCOMES:
Changes in subjective appetite using visual analogue scales | On each test day the appetite questions are answered every 30mins during the 4hour visit.
  Every 30mins, six appetite questions are answered
  * How hungry do you feel?
  * How full do you feel?
  * How strong is your desire to eat?
  * How much do you think you could eat now
  * How thirsty are you?
  * Preoccupation with thoughts of food?
Ad libitum food intake | Recorded at T240mins on the test day visit and then for approximately 12hours at home. Therefore all food consumed during the 24hours of the test day will be assessed
  To assess if each test breakfast provided has an influence on subsequent meals the consumption of the following are recorded:
  - Ad libitum pasta meal: 15% protein; 30% fat and 55% CHO as a homogenous mix and energy density of around 400kJ/100g - served in excess at lunchtime as an individual 600g portion to 'help-yourself'.
  Participants then record all additional meals & snacks consumed at home in a food diary

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Johnstone, Dr, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Institute of Nutrition & Health, University of Aberdeen, Aberdeen, Aberdeen City, United Kingdom

REFERENCES:
- [Background] Bellissimo N, Desantadina MV, Pencharz PB, Berall GB, Thomas SG, Anderson GH. A comparison of short-term appetite and energy intakes in normal weight and obese boys following glucose and whey-protein drinks. Int J Obes (Lond). 2008 Feb;32(2):362-71. doi: 10.1038/sj.ijo.0803709. Epub 2007 Aug 14. PMID 17700578
- [Background] Anderson GH, Tecimer SN, Shah D, Zafar TA. Protein source, quantity, and time of consumption determine the effect of proteins on short-term food intake in young men. J Nutr. 2004 Nov;134(11):3011-5. doi: 10.1093/jn/134.11.3011. PMID 15514267
- [Background] Luhovyy BL, Akhavan T, Anderson GH. Whey proteins in the regulation of food intake and satiety. J Am Coll Nutr. 2007 Dec;26(6):704S-12S. doi: 10.1080/07315724.2007.10719651. PMID 18187437
- [Background] Gustafson DR, McMahon DJ, Morrey J, Nan R. Appetite is not influenced by a unique milk peptide: caseinomacropeptide (CMP). Appetite. 2001 Apr;36(2):157-63. doi: 10.1006/appe.2000.0392. PMID 11237351
- [Background] Burton-Freeman BM. Glycomacropeptide (GMP) is not critical to whey-induced satiety, but may have a unique role in energy intake regulation through cholecystokinin (CCK). Physiol Behav. 2008 Jan 28;93(1-2):379-87. doi: 10.1016/j.physbeh.2007.09.010. Epub 2007 Oct 26. PMID 17964616
- [Background] DiMeglio DP, Mattes RD. Liquid versus solid carbohydrate: effects on food intake and body weight. Int J Obes Relat Metab Disord. 2000 Jun;24(6):794-800. doi: 10.1038/sj.ijo.0801229. PMID 10878689
- [Background] Mattes RD. Beverages and positive energy balance: the menace is the medium. International Journal of Obesity 30: S60-S65, 2006.
- [Background] Wolf A, Bray GA, Popkin BM. A short history of beverages and how our body treats them. Obes Rev. 2008 Mar;9(2):151-64. doi: 10.1111/j.1467-789X.2007.00389.x. PMID 18257753
- [Background] Ludwig DS, Peterson KE, Gortmaker SL. Relation between consumption of sugar-sweetened drinks and childhood obesity: a prospective, observational analysis. Lancet. 2001 Feb 17;357(9255):505-8. doi: 10.1016/S0140-6736(00)04041-1. PMID 11229668
- [Background] Mourao DM, Bressan J, Campbell WW, Mattes RD. Effects of food form on appetite and energy intake in lean and obese young adults. Int J Obes (Lond). 2007 Nov;31(11):1688-95. doi: 10.1038/sj.ijo.0803667. Epub 2007 Jun 19. PMID 17579632
- [Background] Drewnowski A, Bellisle F. Liquid calories, sugar, and body weight. Am J Clin Nutr. 2007 Mar;85(3):651-61. doi: 10.1093/ajcn/85.3.651. PMID 17344485
- [Background] Anderson GH. Much ado about high-fructose corn syrup in beverages: the meat of the matter. Am J Clin Nutr. 2007 Dec;86(6):1577-8. doi: 10.1093/ajcn/86.5.1577. No abstract available. PMID 18065571
- [Background] Kissileff HR, Gruss LP, Thornton J, Jordan HA. The satiating efficiency of foods. Physiol Behav. 1984 Feb;32(2):319-32. doi: 10.1016/0031-9384(84)90147-1. PMID 6718557
- [Background] Kissileff HR. Effects of physical state (liquid-solid) of foods on food intake: procedural and substantive contributions. Am J Clin Nutr. 1985 Nov;42(5 Suppl):956-65. doi: 10.1093/ajcn/42.5.956. PMID 4061368
- [Background] Rolls BJ, Fedoroff IC, Guthrie JF, Laster LJ. Foods with different satiating effects in humans. Appetite. 1990 Oct;15(2):115-26. doi: 10.1016/0195-6663(90)90044-9. PMID 2268137
- [Background] Akhavan T, Luhovyy BL, Anderson GH. Effect of drinking compared with eating sugars or whey protein on short-term appetite and food intake. Int J Obes (Lond). 2011 Apr;35(4):562-9. doi: 10.1038/ijo.2010.163. Epub 2010 Aug 24. PMID 20733582
- [Background] Westerterp-Plantenga MS, Lejeune MP, Nijs I, van Ooijen M, Kovacs EM. High protein intake sustains weight maintenance after body weight loss in humans. Int J Obes Relat Metab Disord. 2004 Jan;28(1):57-64. doi: 10.1038/sj.ijo.0802461. PMID 14710168
- [Background] Weigle DS, Breen PA, Matthys CC, Callahan HS, Meeuws KE, Burden VR, Purnell JQ. A high-protein diet induces sustained reductions in appetite, ad libitum caloric intake, and body weight despite compensatory changes in diurnal plasma leptin and ghrelin concentrations. Am J Clin Nutr. 2005 Jul;82(1):41-8. doi: 10.1093/ajcn.82.1.41. PMID 16002798
- [Background] Lacroix M, Mosora F, Pontus M, Lefebvre P, Luyckz A, Lopez-Habib G. Glucose naturally labeled with carbon-13: use for metabolic studies in man. Science. 1973 Aug 3;181(4098):445-6. doi: 10.1126/science.181.4098.445. PMID 4718109